CLINICAL TRIAL: NCT00387361
Title: Osteopathic Manipulative Treatment (OMT) as Possible Prophylaxis Against Post-Operative Nausea and Vomiting (PONV) in Patients Receiving Inhalational Anesthesia
Brief Title: Osteopathic Manipulative Treatment for Post-Operative Nausea and Vomiting
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of North Texas Health Science Center (Other)
Responsible Party: Hollis H King, DO, PhD, Adjunct Faculty
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2006-56
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Last update posted 2011-01-12 (Estimated); Status verified 2011-01

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Post-Operative Nausea; Nausea; Anesthesia; Osteopathic Manipulative Treatment; Osteopathic Manipulative Medicine; Manipulation, Osteopathic; Osteopathy; Texas College of Osteopathic Medicine
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Nausea | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Procedure: Osteopathic Manipulative Treatment
- 2 (No Intervention)

INTERVENTIONS:
Procedure: Osteopathic Manipulative Treatment — 20 minute post-operative osteopathic manipulation as described in the protocol
  Arms: 1

SUMMARY:
The purpose of this study is to determine if Osteopathic Manipulative Treatment (OMT) is effective in reducing nausea and vomiting experienced by patients recovering from anesthesia. OMT is a treatment in which the physician places his hands on areas of the body and applies pressure to correct disturbances in one area that may be related to a problem in another area of the body. Osteopathic Manipulative Medicine is a specialty for a physician who uses OMT.

The hypothesis of this study is when OMT is combined with standard-of-care prophylactic anti-emetic therapy in patients following administration of inhalational anesthesia, in comparison to a control group receiving only standard-of-care anti-emetic prophylaxis there will be a reduction in the incidence and severity of PONV.

DETAILED DESCRIPTION:
This research study is a prospective, randomized, single-blinded, controlled, clinical trial under the principal investigator, Hollis King, DO, PhD with the University of North Texas - Health Science Center, Texas College of Osteopathic Medicine. The purpose of this study is to determine the effectiveness of osteopathic manipulative treatment (OMT) as an adjunctive modality to standard medical care for reduction of post-operative nausea and vomiting (PONV). This is the first attempt to study the treatment of PONV utilizing OMM; this study is being conducted as a pilot study

The hypothesis of this study is when OMT is combined with standard-of-care prophylactic anti-emetic therapy in patients following administration of inhalational anesthesia, in comparison to a control group receiving only standard-of-care anti-emetic prophylaxis there will be a reduction in the incidence and severity of PONV.

Two aims will guide this study toward evaluation of the hypothesis:

AIM I: To demonstrate the effect of OMT and standard care on the number of episodes of emesis experienced post-operatively by subjects having undergone anesthesia utilizing inhalational anesthesia (alone or in combination with intravenous anesthetics). All subjects will receive the treatment or "no-treat" protocol to which they are randomized. Data will be collected prior to discharge from the post-anesthesia care unit (PACU) to enumerate the episodes of emesis experienced by each study subject. Subjects will be asked to complete the Ambulatory Surgery-Rhodes Index of Nausea, Vomiting, and Retching (AS-RINVR) 24-48 hours following surgery when a post-study questionnaire is completed.1

AIM II: To demonstrate the effect of OMT and standard care on the intensity of nausea experienced post-operatively by subjects having undergone anesthesia utilizing inhalational anesthesia (alone or in combination with intravenous anesthetics). Following a subject's completion of the treatment protocol (or "no-treat" if so randomized), the nausea visual analog scale (VAS) validated by Boogaerts will be employed at 30 minutes, 1 hour, and 24-36 hours following their post-operative, post-anesthesia treatment protocol. Results will be compared between the control and experimental group for differences.

Osteopathic manipulative medicine (OMM) and OMT seek, in general, to facilitate a more optimal and often faster return to health and homeostasis. Though individuals largely seek out OMT for alleviation of structural and musculoskeletal complaints, its uses have been speculated and discovered to have effects also on physiologic mechanisms. Osteopathic manipulative treatment maneuvers to the head, neck, and upper thoracic spine may impart postulated mechanisms for PONV.3 Successful treatment will be measured by the reduction of PONV, as evaluated on several outcome measures, in a group of subjects receiving post-operative OMT along with standard-of-care treatment over those in the control group only receiving standard-of-care treatment for their PONV. Successful completion of all of the above specific aims will not only validate the hypothesis of this study but will also establish the study's effect and feasibility for future study. Additionally, this pilot study will establish the statistical trends needed to establish effect size data which is needed for power analysis and sample size estimates for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Surgery Type: orthopedic surgical procedures of the extremities (including, but not limited to, shoulder, elbow, wrist, hip, knee, and ankle) with estimated blood loss < 250 cc
* Surgery Duration: 30-180 minutes
* Anesthesia Type: General
* Procedure to be conducted at John Peter Smith Hospital
* Age: 18-75
* American Society of Anesthesiologists Classification < 3

Exclusion Criteria:

* Presence or likelihood of joint sepsis
* Confirmed or suspected pregnancy
* *Increased intracranial pressure, skull fracture, or head trauma within 3 months prior to surgery (by history)
* *Oxygen dependence at home (by history)
* *Active or chronic hepatitis B or C (by history)
* *Hepatocellular carcinoma (by history)
* *Disruption of Blood-Brain barrier: uncontrolled HTN, tumor (current or history of), meningitis or encephalitis (within 3 months prior to surgery), epilepsy (by history)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-12; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Reduction in the episodes of emesis
Reduction in the intensity of nausea

SECONDARY OUTCOMES:
Post-anesthesia recollection of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hollis H King, DO, PhD, Principal Investigator — UNTHSC - TCOM, Department of OMM; Osteopathic Research Center; Simon L Schrick-Senasac, OMS-IV, PDF, Study Director — UNTHSC-TCOM, Department of OMM

REFERENCES:
- [Background] Fetzer SJ, Hand MC, Bouchard PA, Smith H, Jenkins MB. Evaluation of the Rhodes Index of Nausea and Vomiting for ambulatory surgery patients. J Adv Nurs. 2004 Jul;47(1):74-80. doi: 10.1111/j.1365-2648.2004.03067.x. PMID 15186470
- [Background] Scuderi PE, Conlay LA. Postoperative nausea and vomiting and outcome. Int Anesthesiol Clin. 2003 Fall;41(4):165-74. doi: 10.1097/00004311-200341040-00012. No abstract available. PMID 14574220
- [Background] Boogaerts JG, Vanacker E, Seidel L, Albert A, Bardiau FM. Assessment of postoperative nausea using a visual analogue scale. Acta Anaesthesiol Scand. 2000 Apr;44(4):470-4. doi: 10.1034/j.1399-6576.2000.440420.x. PMID 10757584
- [Background] Willard FH. Autonomic nervous system. In: Ward, Robert C., D.O., F.A.A.O., ed. Foundations for Osteopathic Medicine. 2nd ed. Philadelphia: Lippincott Williams & Wilkins; 2003:90.
- [Background] American Society of Anesthesiologists. ASA Physical Status Classification System. Available at: http://www.asahq.org/clinical/physicalstatus.htm. Accessed May 11, 2006.
- See also: Website of the American Osteopathic Association — http://www.osteopathic.org